CLINICAL TRIAL: NCT01511705
Title: Open Label, Balanced, Randomized, Two-treatment, Two-period, Two Sequence, Single Dose, Crossover, Oral Bioequivalence Study of Ondansetron Hydrochloride Tablets 8 mg With Zofran® (Containing Ondansetron Hydrochloride Dihydrate) Tablets 8 mg in Healthy, Adult, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study for Ondansetron Hydrochloride Tablets 8 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3873/06-07
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2006-10

CONDITIONS: Healthy
Keywords: Bioequivalence; Ondansetron; crossover
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron Hydrochloride Tablets 8 mg (Experimental): Ondansetron Hydrochloride Tablets 8 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Ondansetron Hydrochloride
- Zofran Tablets 8 mg (Active Comparator): Zofran Tablets 8 mg of GlaxoSmithKline
  Interventions: Drug: Ondansetron Hydrochloride

INTERVENTIONS:
Drug: Ondansetron Hydrochloride — Ondansetron Hydrochloride Tablets 8 mg
  Other Names: Ondansetron Hydrochloride 8 mg (Dr. Reddy's Laboratories)
  Arms: Ondansetron Hydrochloride Tablets 8 mg
Drug: Ondansetron Hydrochloride — Zofran Tablets 8 mg
  Arms: Zofran Tablets 8 mg

SUMMARY:
This is an open label, balanced, randomized, two-treatment, two-period, two sequence,single dose, crossover, oral bioequivalence study.

DETAILED DESCRIPTION:
The study was an open label, balanced, randomized, two-treatment, two-period, two sequence,single dose, crossover, oral bioequivalence study of Ondansetron Hydrochloride tablets 8 mg of Dr. Reddy's Laboratories Limited, India comparing with that of Zofran® (containing Ondansetron Hydrochloride Dihydrate) tablets 8 mg of GlaxoSmithKline, USA in healthy, adult, human subjects under fasting condition. 26 subjects are enrolled in the study, and 24 subjects are completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provide written informed consent.
* Subjects who were healthy adults within 18 and 45 years of age (both inclusive).
* Body mass index of ≥ 18 kg/m2 and ≤ 25 kg/m2, with body weight not less than 50 kg.
* Subjects who had normal health as determined by medical history and physical examination performed within 15 days prior to the dosing of period I.
* Had normal ECG, Chest X-ray and vital signs
* Availability of subjects for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
* If subject is a female volunteer and is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s),such as condoms, foams, jellies, diaphragm, intrauterine device(IUD), or abstinence.

or

* is postmenopausal for at least 1 year or
* is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)
* Each female subject were supposed to undergo a urine pregnancy test to check-in for period-I, period-II and post study.

Exclusion Criteria:

* Subjects incapable of understanding the informed consent.
* Subjects BP ≤ 9060 mm/Hg or BP ≥ 140/90 mm/Hg.
* History of hypersensitivity or idiosyncratic reaction to ondansetron or any other related drugs.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function. Subjects with a history of tuberculosis, epilepsy, asthma(during past 5 years), diabetes, psychosis or glaucoma were not eligible for the study.
* Regular smoker who smokes more than ten cigarettes daily and has difficulty in abstaining from smoking for the duration of each study period.
* Subjects who has taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication with the past 30 days prior to dosing in Period-I.
* History of any psychiatric illness, which may impair the ability to provide written informed consent.
* Subjects who have a history of alcohol or substance abuse within the last 5 years.
* Subjects with clinically significant abnormal values of laboratory parameters.
* Subjects who have participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
* Subjects who are unable to or likely to be non-complaint with protocol requirements or restrictions.
* Any subject in whom ondansetron is contraindicated for medical reasons.
* Subjects who are intolerant to venipuncture.
* Subjects with positive urine screen for drugs of abuse. All subjects urine samples assayed for the presence of drugs of abuse at each study period check-in. Subjects who found to have urine concentrations of any of the tested drugs were not allowed to participate.
* Female volunteers who has used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives with 14 days before dosing.
* Female volunteers who are not negative in pregnancy test
* All female subjects were to be screened for pregnancy at check in of each study period. Subjects with positive or inconclusive results were to be withdrawn from the study.
* Female volunteers who are currently breast feeding.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study were not to be allowed to participate. Female subjects of child bearing potential must either abstain form sexual intercourse or use a reliable barrier method (e.g condom, IUD) or contraception during the course of the study (first dosing until last blood collection) or they were not to be allowed to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Area unde curve (AUC) | First one was within 1 hour prior to drug administration (0.0) and others at 0.33,0.67,1,1.33, 1.67, 2, 2.5, 3, 3.5,4,6,9,12,15,18 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr. I.S Gandhi, Principal Investigator — Vimta Labs Limited
Locations (1):
- Vimta Labs Limited, Hyderabad, Andhra Pradesh, India